CLINICAL TRIAL: NCT02544880
Title: PDE5 Inhibition Via Tadalafil (Cialis®) to Enhance Anti-Tumor MUC1 Vaccine Efficacy in Patients With Resectable, and Recurrent or Second Primary Head and Neck Squamous Cell Carcinoma (HNSCC): A Phase I/II Clinical Trial
Brief Title: PDE5 Inhibition Via Tadalafil to Enhance Anti-Tumor Mucin 1 (MUC1) Vaccine Efficacy in Patients With HNSCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Donald T. Weed, MD, FACS (Other)
Responsible Party: Sponsor-Investigator, Donald T. Weed, MD, FACS, Professor, University of Miami
Organization: University of Miami (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20140960
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer
Keywords: HNSCC; Tadalafil; PDE5 Inhibition; Anti-MUC1 Vaccine; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent HNSCC; Second primary site disease stage III; Second primary site disease stage IV; Anti-Influenza Vaccine
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Tadalafil; poly ICLC; FluBlok

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Tadalafil plus Vaccine Group (Phase I) (Experimental): The first 6 participants will be enrolled in the open label Phase I portion of the study and will receive Tadalafil, Anti-mucin 1 (MUC1) Vaccine and the Anti-Influenza Vaccine for 5 courses. A standard of care (SOC) tumor removal surgery will be completed after the completion of Course 1. Course 2 will resume 5-8 weeks after completion of SOC tumor removal surgery.
  Interventions: Drug: Tadalafil; Biological: Anti-MUC1 Vaccine; Biological: Anti-Influenza Vaccine
- Tadalafil plus Vaccine Group (Phase II) (Experimental): After completion of the Phase I portion of the study, new participants will be enrolled for the randomized, placebo-controlled Phase II. Participants randomized in this group will receive Tadalafil, Anti-MUC1 Vaccine and the Anti-Influenza Vaccine for 5 courses. A standard of care (SOC) tumor removal surgery will be completed after the completion of Course 1. Course 2 will resume 5-8 weeks after completion of SOC tumor removal surgery.
  Interventions: Drug: Tadalafil; Biological: Anti-MUC1 Vaccine; Biological: Anti-Influenza Vaccine
- Tadalafil plus Vaccine Placebo Group (Phase II) (Experimental): After completion of the Phase I portion of the study, new participants will be enrolled for the randomized, placebo-controlled Phase II. Participants randomized in this group will receive Tadalafil, placebo for the Anti-MUC1 Vaccine and placebo for the Anti-Influenza Vaccine for 5 courses. A standard of care (SOC) tumor removal surgery will be completed after the completion of Course 1. Course 2 will resume 5-8 weeks after completion of SOC tumor removal surgery.
  Interventions: Drug: Tadalafil; Other: Anti-MUC1 Vaccine Placebo; Other: Anti-Influenza Vaccine Placebo
- Tadalafil Placebo plus Vaccine Group (Phase II) (Experimental): After completion of the Phase I portion of the study, new participants will be enrolled for the randomized, placebo-controlled Phase II. Participants randomized in this group will receive placebo for Tadalafil, the Anti-MUC1 Vaccine and the Anti-Influenza Vaccine for 5 courses. A standard of care (SOC) tumor removal surgery will be completed after the completion of Course 1. Course 2 will resume 5-8 weeks after completion of SOC tumor removal surgery.
  Interventions: Biological: Anti-MUC1 Vaccine; Biological: Anti-Influenza Vaccine; Other: Tadalafil Placebo
- Control Group (Other): For eligible participants who opt out of receiving study intervention. Participants in this group will receive SOC treatment only.
  Interventions: Other: Standard of Care Treatment

INTERVENTIONS:
Drug: Tadalafil — Tadalafil tablets administered by mouth. Dose will be between 10 to 20 mg adjusted depending on patient's body weight. On course 1, Tadalafil will be administered daily for 19 consecutive days. On Course 2 through 4, Tadalafil will be administered daily for 14 consecutive days. No Tadalafil will be provided on Course 5.
  Other Names: Cialis
  Arms: Tadalafil plus Vaccine Group (Phase I); Tadalafil plus Vaccine Group (Phase II); Tadalafil plus Vaccine Placebo Group (Phase II)
Biological: Anti-MUC1 Vaccine — 300 uL Anti-MUC1 vaccine will be administered intramuscularly in the right upper limb. Anti-MUC1 vaccine will be administer on Day 7 on course 1, on Day 10 for courses 2 through 4 and on Day 1 on course 5.
  Other Names: Hiltonol
  Arms: Tadalafil Placebo plus Vaccine Group (Phase II); Tadalafil plus Vaccine Group (Phase I); Tadalafil plus Vaccine Group (Phase II)
Biological: Anti-Influenza Vaccine — 300 uL Anti-Influenza vaccine will be administered intramuscularly in the left upper limb. Anti-Influenza vaccine will be administer on Day 7 on course 1, on Day 10 for courses 2 through 4 and on Day 1 on course 5.
  Other Names: Flublok
  Arms: Tadalafil Placebo plus Vaccine Group (Phase II); Tadalafil plus Vaccine Group (Phase I); Tadalafil plus Vaccine Group (Phase II)
Other: Tadalafil Placebo — Placebo tablets mimicking Tadalafil administered by mouth. On course 1, Tadalafil Placebo will be administered daily for 19 consecutive days. On Course 2 through 4, Tadalafil placebo will be administered daily for 14 consecutive days. No Tadalafil Placebo will be provided on Course 5.
  Arms: Tadalafil Placebo plus Vaccine Group (Phase II)
Other: Anti-MUC1 Vaccine Placebo — Placebo for Anti-MUC1 vaccine will be administered intramuscularly in the right upper limb. Placebo for Anti-MUC1 vaccine will be administer on Day 7 on course 1, on Day 10 for courses 2 through 4 and on Day 1 on course 5..
  Arms: Tadalafil plus Vaccine Placebo Group (Phase II)
Other: Standard of Care Treatment — Treatment according to prescribed standard of care regimen.
  Arms: Control Group
Other: Anti-Influenza Vaccine Placebo — Placebo for Anti-Influenza vaccine will be administered intramuscularly in the left upper limb. Placebo for Anti-Influenza vaccine will be administer on Day 7 on course 1, on Day 10 for courses 2 through 4 and on Day 1 on course 5.
  Arms: Tadalafil plus Vaccine Placebo Group (Phase II)

SUMMARY:
The investigators hypothesize that Tadalafil treatment, by lowering Myeloid Derived Suppressor Cells (MDSCs) and regulatory T cells (Tregs), can prime an antitumor immune response and promote a permissive environment that should increase the efficacy of anti-tumor vaccine in a setting of minimal residual disease.

DETAILED DESCRIPTION:
This study is halting accrual at the end of the phase 1 portion of the study as data from the phase I study suggest that an alternative approach for the phase 2 portion of the study be undertaken. A newly designed Phase II trial is being developed and will be submitted as a new study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven recurrent or second primary HNSCC of the oral cavity, oropharynx, hypopharynx or larynx (second primary includes unknown primary)
2. Stage III or IV (AJCC, 7th ed., 2010) recurrent or second primary HNSCC (For recurrent tumors, staging is determined by the recurrent stage, not by the original pretreatment stage.)
3. Surgically resectable, recurrent or second primary HNSCC
4. Prior radiation, with or without prior surgery and/or chemotherapy, to the head and neck for definitive treatment of HNSCC of the oral cavity, oropharynx, hypopharynx or larynx with previously documented complete clinical or radiographic response to initial treatment

   * a. Prior radiation and any chemotherapy, must have been completed >4 months prior to biopsy-proven recurrence or second primary site disease
   * b. Recurrent or second primary HNSCC arises within the previously irradiated field
5. Age ≥ 18 years
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2 or equivalent scale score. See Appendix D for equivalent scale criteria.
7. Acceptable organ function as defined by all of the following:

   * Alkaline phosphatase < 4.0 x upper limit of normal (ULN)
   * Aspartate transaminase (AST) ≤ 2.5 x ULN
   * Alanine transaminase (ALT) ≤ 2.5 x ULN
   * calculated Creatinine Clearance ≥ 51ml/min as determined by the Cockcroft-Gault Equation:

     * [(140-age) * (Weight in kg) * (0.85, if female)] / (72 * Cr)
8. Suitable venous access to allow for all study related blood sampling (safety and research)
9. Ability to understand and willingness to sign the written informed consent and Health Insurance Portability and Accountability Act (HIPAA) document/s.

Inclusion Criteria (non-randomized control)

1. Biopsy-proven recurrent or second primary HNSCC of the oral cavity, oropharynx, hypopharynx or larynx (second primary includes unknown primary)
2. Stage III or IV (AJCC, 7th ed., 2010) recurrent or second primary HNSCC (For recurrent tumors, staging is determined by the recurrent stage, not by the original pretreatment stage.)
3. Surgically resectable, recurrent or second primary HNSCC
4. Prior radiation with or without prior surgery and/or chemotherapy, to the head and neck for definitive treatment of HNSCC of the oral cavity, oropharynx, hypopharynx or larynx with previously documented complete clinical or radiographic response to initial treatment

   * a. Prior radiation and any chemotherapy, must have been completed >4 months prior to biopsy-proven recurrence or second primary site disease
   * b. Recurrent or second primary HNSCC arises within the previously irradiated field
5. Age ≥18 years
6. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1 or 2 or equivalent scale score.
7. Suitable venous access to allow for all study related blood sampling (safety and research)
8. Ability to understand and willingness to sign the written informed consent and HIPAA document/s.

Exclusion Criteria:

1. Salvage surgery is not recommended as per National Comprehensive Cancer Network (NCCN) guidelines, or after multidisciplinary treatment evaluation, including those with surgically unresectable disease at primary site or regional lymph nodes
2. Recurrent or second primary AJCC Stage I or II HNSCC (for recurrent tumors, staging is determined by the recurrent stage, not by the original pretreatment stage).
3. Distant metastatic disease
4. Recurrent or second primary HNSCC of the nasopharynx, paranasal sinuses, or cervical esophagus
5. Use of Phosphodiesterase Type 5 (PDE5) inhibitors such as vardenafil (Levitra®), Tadalafil (Cialis®), and sildenafil citrate (Viagra®) ≤15-days prior to (intended) enrollment
6. Patients who have the intention to receive non-study PDE5 inhibitors and flu vaccination(s) anytime during the study will be excluded.
7. Prior or known adverse reactions to PDE5 inhibitors, poly-ICLC (Hiltonol®), and prior dose(s) of Influenza vaccine including but not limited to their components
8. History of severe or unstable cardiac or cerebrovascular disease:

   * a. Myocardial infarction within the last 90 days
   * b. Unstable angina or angina occurring during sexual intercourse
   * c. New York Heart Association (NYHA) Class 2 or greater heart failure in the last 3 months.
   * d. Uncontrolled arrhythmias
   * e. Sustained hypotension (<90/50 mmHg) or uncontrolled Hypertension (>170/100 mmHg)
   * f. Stroke within the last 6 months
9. Therapy with nitrates, alpha-blockers, or cytochrome P450 (CYP3A4) inhibitors within 7-days prior to study treatment initiation and for whom stopping is unsafe and/or a safe substitute is not medically recommended. Some examples are provided in Appendix A.
10. Positive Antinuclear Antibody Test (ANA)
11. Immunosuppression or immunocompromised for reasons not directly related to patient's malignancy (e.g. HIV or kidney transplant)
12. History of severe or life threatening autoimmune diseases [Exceptions: Mild autoimmune diseases determined at the discretion of the Investigator(s), e.g. psoriasis.]
13. Unilateral blindness, hereditary retinal disorders, or at an increased risk of blindness
14. Unilateral deafness, or severe hearing loss dependent upon hearing aid(s) for serviceable communication
15. Female patients who are pregnant or breastfeeding. (Females of childbearing potential are required to have a negative urine β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women.)
16. Females of childbearing potential who refuse to practice effective methods of contraception or abstain from heterosexual intercourse from the time of signing the informed consent through 30-days after the last vaccination.
17. Serious medical or psychiatric illness/condition, including alcohol or drug abuse likely in the judgment of the Investigator(s) to interfere with compliance to protocol treatment/research.
18. Patients of vulnerable populations such as children less than 18 years of age, prisoners, institutionalized individuals or others likely to be vulnerable are not eligible for participation in this study.

Exclusion Criteria (non-randomized control)

1. Salvage surgery is not recommended as per NCCN guidelines, or after multidisciplinary treatment evaluation, including those with surgically unresectable disease at primary site or regional lymph nodes
2. Recurrent or second primary AJCC Stage I or II HNSCC (for recurrent tumors, staging is determined by the recurrent stage, not by the original pretreatment stage).
3. Distant metastatic disease
4. Recurrent or second primary HNSCC of the nasopharynx, paranasal sinuses, or cervical esophagus
5. Use of PDE5 inhibitors such as vardenafil (Levitra®), Tadalafil (Cialis®), and sildenafil citrate (Viagra®) ≤15-days prior to (intended) enrollment
6. Patients who have the intention to receive non-study PDE5 inhibitors and flu vaccination(s) anytime during the study will be excluded.
7. Positive Antinuclear Antibody Test (ANA)
8. Immunosuppression or immunocompromised for reasons not directly related to patient's malignancy (e.g. HIV or kidney transplant)
9. History of severe or life threatening autoimmune diseases [Exceptions: Mild autoimmune diseases determined at the discretion of the Investigator(s), e.g. psoriasis.]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-04-25 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Phase 1 - Number of participants experiencing adverse events and/or treatment limiting-toxicities after receiving protocol therapy. | Up to 2 Years
  The primary objective of the lead-in, open-label, single-arm, phase I part of study will evaluate the safety of Tadalafil in combination with anti-MUC1/anti-influenza vaccines (TV) in terms of adverse events (AEs), serious adverse events (SAEs) and treatment-limiting toxicities (TLTs).
Phase 2 - Rate of tumor-specific immune response to protocol therapy. | Up to 3.5 years
  The primary objective of phase II is to evaluate immune response (tumor-specific immune response of the anti- MUC1 and anti-influenza vaccines when combined with Tadalafil. Immune response will be evaluated by determining patients' immunological profile (e.g. peripheral blood mononuclear cells (PBMCs), leukocyte subsets, and serum cytokine levels) and immunological reactivity (e.g. through DTH skin test, T cell proliferation, by Enzyme-Linked ImmunoSpot (ELISPOT), specific Immunoglobulin G (IgG) concentration, and immune response by peripheral blood sera) before and after surgery, and during treatment with Tadalafil and the anti-MUC1 and anti-Influenza vaccines.

SECONDARY OUTCOMES:
Phase 1 - Rate of tumor-specific immune response to protocol therapy. | Up to 2 years
  Immune response will be evaluated by determining patients' immunological profile (e.g. peripheral blood mononuclear cells (PBMCs), leukocyte subsets, and serum cytokine levels) and immunological reactivity (e.g. through DTH skin test, T cell proliferation, by ELISPOT, specific IgG concentration, and immune response by peripheral blood sera) before and after surgery, and during treatment with Tadalafil and the anti-MUC1 and anti-Influenza vaccines.
Phase 1/2 - Rate of recurrence-free survival (RFS) in participants | Up to 3.5 years
  The rate of recurrence-free survival (RFS) in patients with recurrent or second primary HNSCC after salvage surgery. RFS is defined as the time from date of Surgery to the date of first documented recurrence. All patients will be rendered disease free (i.e. no measurable disease) after surgery, thus any confirmed evidence of disease recurrence regardless of size or site will constitute the recurrence time point. Recurrence will be demonstrated by clinical assessments such as clinical examinations and tumor assessments (possibly) by CT, PET/CT or MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Donald T Weed, MD, FACS, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weed DT, Zilio S, Reis IM, Sargi Z, Abouyared M, Gomez-Fernandez CR, Civantos FJ, Rodriguez CP, Serafini P. The Reversal of Immune Exclusion Mediated by Tadalafil and an Anti-tumor Vaccine Also Induces PDL1 Upregulation in Recurrent Head and Neck Squamous Cell Carcinoma: Interim Analysis of a Phase I Clinical Trial. Front Immunol. 2019 May 31;10:1206. doi: 10.3389/fimmu.2019.01206. eCollection 2019. PMID 31214178
- See also: The Reversal of Immune Exclusion Mediated by Tadalafil and an Anti-tumor Vaccine Also Induces PDL1 Upregulation in Recurrent Head and Neck Squamous Cell Carcinoma: Interim Analysis of a Phase I Clinical Trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6554471/